CLINICAL TRIAL: NCT03522636
Title: Effect of Pre-hospital Blood Transfusion on Early Outcomes in Trauma Patients Transported by Physician-staffed HEMS (Helicopter Emergency Medical Service)
Brief Title: Rapid Administration of Blood by HEMS in Trauma
Acronym: RABBIT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zdravotnicka Zachranna Sluzba Kralovehradeckeho Kraje (Other)
Collaborators: University Hospital Hradec Kralove (Other)
Responsible Party: Principal Investigator, Anatolij Truhlar, MD, PhD, FERC, Medical Director EMS, Zdravotnicka Zachranna Sluzba Kralovehradeckeho Kraje
Other Study IDs: 20180001
Record Dates: First submitted 2018-03-31; First posted 2018-05-11 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Wounds and Injuries; Acute Coagulopathy; Trauma
Keywords: Prehospital transfusion; Trauma; Trauma induced coagulopathy
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment: Prehospital blood products resuscitation up to 2 units of blood products as follows: 1 unit of packed human plasma and 1 unit of packed red blood cells
- Historic control: No prehospital blood products available

SUMMARY:
Trauma is a leading cause of death among people younger than 44 years. Five million people worldwide die from trauma annually. Uncontrolled haemorrhage causing traumatic-haemorrhagic shock (THS) is the leading cause of potentially preventable deaths from severe trauma. Uncorrected hypervolaemia and prolonged shock cause severe tissue hypoperfusion, vital organ ischemia and subsequently acidosis. In up to one third of trauma patients, laboratory findings suggest traumatic induced coagulopathy, which is further triggered by loss or dilution of coagulation factors. These patients have a significantly increased morbidity and mortality compared to patients with similar injury patterns without coagulopathy. Minimizing the time to surgical control of haemorrhage is key in order to improve outcome. However, immediate and goal directed volume and coagulation resuscitation including use of blood transfusion is crucial to enable survival until definitive hospital care. The primary objective of this study will be to evaluate feasibility of prehospital administration of 1 unit of human plasma and 1 unit of red blood cells, and explore association of early prehospital transfusion with early outcomes in patients presenting with THS, severe bleeding or peri-arrest state who are matching indication criteria and are transported by Helicopter Emergency Medical Service. Results of clinical examinations and laboratory variables in a group of patients receiving prehospital transfusion will be compared to matched population of patients treated before blood has been available on board. Secondary aim of the study is to detect any potential logistical and/or organisational adverse effects, incl. cost-effectiveness, in a regional trauma system with prehospital times (time of injury to trauma centre) ranging from 45 to 75 minutes.

DETAILED DESCRIPTION:
Background and rationale of the project Trauma is a leading cause of death among people younger than 44 years. Uncontrolled haemorrhage causing traumatic-haemorrhagic shock (THS) is the leading cause of potentially preventable deaths from severe trauma. Uncorrected hypervolaemia and prolonged shock cause severe tissue hypoperfusion, vital organ ischemia and subsequently acidosis. Shock, acidosis and hypothermia are recognized drivers of anti-coagulant and fibrinolytic pathways. In up to one third of trauma patients, laboratory findings suggest traumatic induced coagulopathy, which is further triggered by loss or dilution of coagulation factors. These patients have a significantly increased morbidity and mortality compared to patients with similar injury patterns without coagulopathy. Minimizing the time to surgical control of haemorrhage is key in order to improve outcome. However, immediate and goal directed volume and coagulation resuscitation including use of blood product transfusion is crucial to enable survival until definitive hospital care.

Role of HEMS in a trauma system. Helicopter Emergency Medical Services (HEMS) can rapidly deliver advanced medical care and speed up patient transport to designated trauma centres. In the Czech Republic, HEMS covers 76.5% of the area and 99.4% of the population of the Czech Republic within 20 minutes since the emergency call is received via Emergency Medical Dispatch Centre (EMDC). HEMS Hradec Kralove is one of the well-recognized systems in the country. Its catchment area is 1.1 million inhabitants living in the Hradec Kralove and Pardubice regions. Trauma patients include 100-120 multiple trauma injuries and 50-60 isolated traumatic brain injuries (TBI) annually. In 2017, there were 95.9% primary flights (to the scene of accident), of which 81.9% take-offs were decided by EMDC dispatchers immediately after receiving an emergency call. Management of patients in THS requires early identification of the bleeding source, use of effective techniques to stop compressible haemorrhage, support of clot formation and minimisation of on-going blood loss in non-compressible haemorrhage, judicious fluid resuscitation with monitoring of effect, and a pre-alert system for damage control resuscitation or surgery at the receiving hospital. HEMS teams must be skilled to recognise and treat massive bleeding and acute traumatic coagulopathy in the pre-hospital environment.

Diagnostics of THS. Haemorrhage leads to a fall in systemic filling pressure and venous return. The resulting decrease in cardiac minute volume, and therefore in oxygen and nutrient supply, sets off an endogenous stress response aiming to maintain perfusion pressure. Thus, blood pressure and heart rate must be interpreted with caution, and cardiac output might have dropped to some 60% until blood pressure will start to decrease. Although a systolic blood pressure <90 mmHg is the typically considered as the leading symptom of hypovolemic shock, clinical assessment of trauma patients comprises on-going and repeated evaluation of the mental status, capillary filling time, clinical appearance, changes in heart rate, and mechanism of injury. Current literature suggests that the combined evaluation of heart rate, SABP, Glasgow Coma Scale (GCS) and the ability to maintain a patent airway increases the predictability for advanced in-hospital interventions up to four times. This is of particular importance for an in-hospital blood transfusion request policy. Suitable triggers for preparation for massive transfusion are suspicion or evidence of active haemorrhage, incl. trauma triage criteria, systolic arterial blood pressure (SABP) < 90 mmHg, failure to respond to a fluid bolus, heart rate > 120/min, and penetrating injuries. Accordingly, physical examination on scene should focus on injury patterns known to cause haemorrhage such as penetrating trauma, pelvic or femoral fractures and blunt abdominal trauma.

Prehospital treatment of THS. The up-to-date concept of initial trauma care is called damage control resuscitation, which comprises hypotensive resuscitation, haemostatic resuscitation and damage control surgery. Control of haemorrhage is crucial in order to interrupt the vicious circle of blood loss, hypervolaemia, hypoperfusion, acidosis and coagulopathy, finally resulting in therapy refractory shock and death. Basic techniques like direct compression, pressure dressings, tourniquets, traction devices and pelvic splints are used routinely in obvious or suspicious bleeding. In life threatening haemorrhagic shock, fluid resuscitation is still the main stem therapy. The primary and ultimate goal of pre-hospital fluid resuscitation is to prevent hypovolemic cardiac arrest and to minimize organ damage caused by prolonged or uncorrected hypotension causing organ ischemia. For this reason permissive hypotension should only be applied in the first hour after the insult. There are extensive side effects of fluid resuscitation in uncontrolled bleeding patients. Inappropriate or over-infusion has been shown to harm and to worsen outcome. Hypotensive resuscitation is a temporary strategy for management of patients with uncontrolled blood loss until the source of bleeding is controlled. Fluid resuscitation should be spared or postponed in patients with uncontrolled haemorrhage, normal mental status and SABP > 90 mmHg. Fluids should be titrated in uncontrolled bleeding patients without head trauma to a target SABP around 90 mmHg. However, it is noteworthy that the concept of hypotensive resuscitation must be tailored and adjusted to the patients need. In patients with severe traumatic brain injury higher SABP must be achieved with higher amounts of fluids and very seldom use of vasopressor drugs when necessary. There is an on-going debate which fluids and what amounts should be considered optimal for haemorrhagic shock management. Colloids did not show to improve outcome when compared with crystalloids. The same is true for hyperosmolar solutions. Compared to the United Kingdom, Scandinavia and other highly developed countries, there are no prehospital blood products currently available in Central, Southern and Eastern Europe, partially because of high logistic and material demands, risk of wasting, high expenses, and unproven benefit of prehospital use of red blood cells without plasma.

Co-operation between HEMS and a trauma centre. The regional trauma system in the Hradec Kralove Region has been gradually developed during last couple of years. One of its main advantages is excellent long-term co-operation between EMDC, HEMS, and receiving trauma centre, incl. quality management. There are different triage tools used to help to outline patient routes to trauma centres. These latter can include immediate need for blood or life saving surgery. In Hradec Kralove, it was for the first time in the Czech Republic, when a new concept of trauma triage was implemented and improved on-scene triage. The triage criteria were adopted from the American College of Surgeons (ACS) and include: mechanism of injury (e.g. fall from height > 6 m, person trapped in a vehicle), anatomical and physiological criteria, and selected special considerations (e.g. age, comorbidities). Its specificity is 8-10% and sensitivity 95-97%. The same triage system was later implemented into all other prehospital systems, integrated into the nation-wide recommendations of the Ministry of Health (Trauma Care in the Czech Republic) and Guidelines of the Czech Society for Emergency and Disaster Medicine ČLS JEP. Use of pre-hospital triage can predict risk of THS and need for specialized trauma care.

Prehospital blood transfusion. Haemostatic resuscitation is the very early use of blood products as primary resuscitation fluid to prevent exsanguination by trauma-induced coagulopathy. The recommended ratio of packed red cells, fresh frozen plasma and platelets is 1:1:1. In a few locations around the world, physician led HEMS teams provide advanced medical interventions such as thoracotomy, resuscitative endovascular balloon occlusion of aorta (REBOA), and blood product (BP) transfusion which traditionally occurred in the highly specialized hospital centres. Administration of BPs in a helicopter has been studied in specific cohorts including either longer transport times to definitive treatment facility, high prevalence of penetrating thorax and epigastrium injuries, or war injuries with restricted medical care. The potential role of packed red blood cells is yet to be identified, although many HEMS systems already demonstrated feasibility. Recent systematic review searching bibliographic databases to July 2015 did not identify any prospective comparative or randomized studies on prehopsital use of BPs. A single study showed improved survival in the first 24 hours, but vast majority of studies provided very low quality of evidence. None of these studies was performed on a cohort of patients similar to the population treated in our setting: blunt injuries and short prehospital times. Transfusion reactions were rare, suggesting the short-term safety of prehospital BP administration equal to those occurring at emergency departments. Current practice at the HEMS Hradec Kralove is to prealert the admitting facility and request blood products from the scene. These are available after helicopter arrival at hospital. It was calculated that availability of BPs on board would result in earlier BP transfusion for at least 20-30 minutes compared to current situation.

Hypothesis. Given evidence in support of massive transfusion protocol in hospitals, the investigators hypothesize that early prehospital BP transfusion will be associated with lower risk of THS and coagulopathy on admission to the trauma centre, and during 24 hours after admission. Lower requirements for BP transfusion during 24 hours after admission, improved 24-hour mortality, and outcome on discharge from hospital are also expected.

Statistical analysis. Conditional logistic regression and mixed-effects linear regression will be used to determine the association of early administration of BP transfusion with outcome variables. Patients receiving BP transfusion are supposed to be more severely injured with a higher risk of mortality. Because of this, we cannot compare their outcome data to those of patients without prehospital BP transfusions, but with a retrospective cohort of patients who had received massive transfusion protocol already requested by HEMS from the scene during the period of previous 12/24 months before implementation of BP transfusion into HEMS. To prevent selection bias, the propensity score model will be developed to predict the likelihood of receiving BP transfusion based on several prehospital variables to allow appropriate matching of treated and control patients based on this probability of receiving BP transfusion. Covariates in the propensity score model will include age, SABP, heart rate, crystalloid volume before HEMS arrival (if given by a ground ambulance team), crystalloid volume during HEMS transport, type of injury (blunt vs. penetrating), prehospital time and distance to hospital. Covariates for 24-hour survival will include at least sex, Injury Severity Score (ISS), SABP, heart rate and Glasgow Coma Score (GCS) at admission, INR, rotational thromboelastometry (ROTEM) parameters (e.g. clotting time, alfa-angle), intensive care unit admission, days of mechanical ventilation, and need for surgery. Similar covariates will be used for THS and trauma induced coagulopathy indicators. Subgroup analysis will be performed for patients with traumatic cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

1. Physiological indications

   1. Hypotension with absent radial pulse
   2. Hypotension with systolic arterial blood pressure < 100 mmHg
2. Anatomical indications

   1. Penetrating thoracic and/or abdominal injuries with signs of severe bleeding
   2. Injuries to neck, groins and/or axilla with signs of severe bleeding
   3. Clinical signs of intraabdominal bleeding
   4. Unstable chest wall
   5. Unstable pelvis
   6. Closed and/or open fractures of two or more long bones (femur, tibia, humerus)
   7. Open fracture of at least one femur type OIII
   8. Open fracture of pelvis
   9. Partial and/or total amputation limb injury above knee and/or elbow with severe external blood loss
3. Mechanism of injury (supporting indications)

   1. Human torso entrapped in the vehicle with need for extrication (thorax, abdomen, pelvis)
   2. Fall from height of > 6 metres (on scene verification needed)
   3. Human torso (thorax, abdomen, pelvis) over-driven by a motor vehicle
   4. Human torso (thorax, abdomen, pelvis) compressed by a heavy object or animal

Exclusion Criteria:

1. Absolute contraindications

   a. Traumatic cardiac arrest (TCA) from a blunt injury before decision to administer blood products. Any ROSC after resuscitation of TCA is not a contraindication.
2. Relative contraindications

   1. Traumatic brain injury (TBI) caused by direct force towards head region (e.g. gunshot) without signs of injury to other systems or body areas
   2. Age under 15 years.
   3. Any other admitting hospital than trauma center of the University Hospital Hradec Kralove

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All injured patients treated by a physician-staffed HEMS team will be eligible for inclusion. Authorized on-scene HEMS physicians will be responsible to make decision to administer prehospital blood if one or more of the anatomical and/or physiological inclusion criteria are met. Prehospital transfusion will always be considered as a life-saving intervention.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-05-31 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Units of blood products used | Time of injury to 24 hours
  Transfusion units of red blood cells, plasma and platelets

SECONDARY OUTCOMES:
Prehospital time | Time of injury to 24 hours
  Prehospital time (time of injury to arrival at trauma centre)
Volume of pre-hospital fluids | Time of injury to 24 hours
  Volume of fluids (crystalloids) given until hospital admission
Blood pressure on admission to trauma centre | Time of injury to 24 hours
  Systolic and diastolic blood pressure on admission to trauma centre
Trauma-induced coagulopathy | Time of injury to 24 hours
  NR > 1.5 and coagulation variables measured viscoelastically by rotational thromboelastometry (ROTEM)
Lactate concentration | Admission to 24 hours
  Venous lactate concentration
ICU stay | Admission to discharge from acute care hospital or 1 month
  Days of stay at intensive care unit
Days of mechanical ventillation | Time of injury to discharge from acute care hospital or 1 month
  Days of mechanical ventillation
Sepsis-related organ failure assessment (SOFA) score | Admission to discharge from acute care hospital or 1 month
  Sepsis-related organ failure assessment (SOFA) score is based on six different scores, one each for the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems assisting in estimating the risk of morbidity and mortality
Complications | Time of injury to discharge from acute care hospital or 1 month
  Transfusion related reactions, logistical, and organisational complications
24 hour and 30 day mortality | 24 hours and 1 month
  Trauma-related mortality between time of injury and up to discharge from acute care hospital or 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Anatolij Truhlar, MD PhD FERC, Principal Investigator — Zdravotnicka Zachranna Sluzba Kralovehradeckeho Kraje
Locations (2):
- Czechia (2):
  - University Hospital Hradec Kralove, Hradec Králové
  - Zdravotnicka zachranna sluzba Kralovehradeckeho kraje, Hradec Králové